CLINICAL TRIAL: NCT01468142
Title: Pulmonary Pathophysiology and Inflammatory Response in Patients Treated With Ecmo for Severe Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Bernhard Holzgraefe, Consultant, ECMO centre Karolinska, Principal Investigator, Karolinska University Hospital
Other Study IDs: 2011/1282-31/1
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Respiratory Distress Syndrome, Adult; Respiratory Distress Syndrome, Child
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is the observation of the course of

* the mechanics of the respiratory system
* the endexpiratory lung volume
* and the inflammatory response in patients undergoing treatment with extracorporeal life support (ECLS) due to severe refractory respiratory failure at our department.

ELIGIBILITY:
Inclusion Criteria:

* patients accepted for extracorporeal life support at our department due to the most severe forms of ARDS/respiratory failure not responding to conventional therapy.

Exclusion Criteria:

* malignant disease with a poor prognosis
* massive intracranial bleeding

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General hospitals, district hospitals, specialized hospitals,
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Course of inflammatory parameters and lung function | end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Holzgraefe, MD, Principal Investigator — Karolinska University Hospital; Anders Larsson, PhD, Study Chair — Uppsala University, Uppsala, Sweden
Locations (1):
- ECMO Centre Karolinska, Solna, Stockholm County, Sweden